CLINICAL TRIAL: NCT01786460
Title: Brain Injury Biomarkers in the General Population
Status: Completed | Type: Observational
Sponsor: Banyan Biomarkers, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ATO-05
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteers
  Interventions: Other: Blood draw at Days 0, 7, 14, and 21

INTERVENTIONS:
Other: Blood draw at Days 0, 7, 14, and 21

SUMMARY:
The purpose of this study is to use an investigational assay to assess levels of putative biomarkers of traumatic brain injury (TBI) in a general population. The data will be used in a correlative analysis with data collected under a separate study of severe TBI.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and no more than 80 years of age
* Willing to undergo consent
* PI believes volunteer is appropriate candidate for study

Exclusion Criteria:

* Participating in another clinical study that may affect the results of either study
* Non-English speaking
* Venipuncture not feasible
* Blood donation within 1 week of screening
* PI determines volunteer is not medically suitable for study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers who meet eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Assessment of the putative biomarkers for TBI markers in general population using an investigational assay | up to 21 days

SECONDARY OUTCOMES:
Correlation of the putative biomarkers for TBI levels in general population to levels in patients with severe TBI | 0, 14, 7, and 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Jackson Streeter, MD, Study Chair — Banyan Biomarkers
Locations (5):
- United States (5):
  - Office of Nagi S. Ibrahim, Vista, California
  - Shands at University Florida Gainesville, Gainesville, Florida
  - Dekalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - New England Center for Clinical Research, Fall River, Massachusetts